CLINICAL TRIAL: NCT00190801
Title: Open-Label Single-Arm Phase 2 Study of ALIMTA Plus Cisplatin in Korean Patients With Advanced Gastric Carcinoma
Brief Title: Phase 2 Study on Use of a Combination of Pemetrexed in Patients With Advanced Gastric Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6154; H3E-KL-JMFK
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Pemetrexed; Cisplatin

INTERVENTIONS:
Drug: pemetrexed
Drug: cisplatin

SUMMARY:
Pemetrexed has shown an anti-tumor activity in advanced gastric cancer patients in a previous study, while cisplatin is widely used in the combination chemotherapy of gastric cancer. Pemetrexed has shown synergy with cisplatin in preclinical models and in various human cancers. The introduction of vitamin supplementation has made treatment with pemetrexed plus cisplatin safe and well tolerated. The present phase 2 study is an effort to determine the efficacy and safety of the combination of pemetrexed and cisplatin in Korean patients with gastric carcinoma who had no prior palliative chemotherapy for advanced disease. The patients, who will give their consent for participating in this study, will be screened for their eligibility and on meeting pre-defined study eligibility criteria, they will receive an intravenous therapy of the combination of pemetrexed and cisplatin for number of times that in the opinion of their treating physician is appropriate for them. A response rate of 30% is considered as the minimum activity level of interest for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of adenocarcinoma of the stomach
* Stage IV disease not amenable to curative surgery.
* Disease status must be that of measurable disease as defined by RECIST criteria
* Performance Status of 0 or 1 on the ECOG Scale and adequate organ function.
* Signed informed consent from patient

Exclusion Criteria:

* Prior palliative chemotherapy for advanced disease.
* Known or suspected brain metastasis or Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Concurrent administration of any other tumor therapy
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of ALIMTA plus cisplatin.
* Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-09; Study Completion 2005-09

PRIMARY OUTCOMES:
Response rate according to RECIST criteria

SECONDARY OUTCOMES:
The following time to event efficacy measures:
o Duration of overall response for responding patients
o Time to documented progressive disease
o Time to treatment failure
o Overall survival
The quantitative and qualitative toxicity of pemetrexed plus cisplatin in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul